CLINICAL TRIAL: NCT01445249
Title: A Randomised, Blinded Comparison of a Nerve Stimulator Guided Ankle Block Compared to a Landmark Guided Ankle Block for Pain Relief After Forefoot Surgery.
Brief Title: Medial Forefoot Block for Analgesia After Foot Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07/H1304/118
Record Dates: First submitted 2011-08-17; First posted 2011-10-03 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Hallux Valgus
Keywords: regional anaesthetic techniques; surgery orthopaedic
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Landmark guided ankle block (Active Comparator): This group will receive a landmark guided ankle block.
  Interventions: Procedure: Landmark guided ankle block.
- This group will be given a PNS guided ankle block (Active Comparator): Peripheral nerve stimulation will be used in this group to guide local anaesthetic infiltration. The technique is termed medial forefoot block.
  Interventions: Procedure: PNS guided block.

INTERVENTIONS:
Procedure: Landmark guided ankle block. — 25-30mls 0.5% levobupivacaine will be infiltrated to provide a landmark guided ankle block.
  Other Names: Other names not required
  Arms: Landmark guided ankle block
Procedure: PNS guided block. — This group will have 25-30mls of 0.5% levobupivacaine infiltrated as directed by peripheral nerve stimulation.
  Other Names: Other names not required
  Arms: This group will be given a PNS guided ankle block

SUMMARY:
Forefoot surgery includes bunion surgery and similar reconstructive bone cutting surgery and is very painful. Local anaesthetic nerve blocks are used to provide pain relief after this work. The purpose of this study is to compare two techniques: one using anatomical landmarks alone to guide local anaesthetic infiltration, the other using peripheral nerve stimulation to guide local anaesthetic infiltration (termed medial forefoot block). The two techniques will be compared for reliability of postoperative analgesia.

DETAILED DESCRIPTION:
More extensive description not desired.

ELIGIBILITY:
Inclusion Criteria:

* Fit adults requiring forefoot surgery with bone cutting

Exclusion Criteria:

* Morbid obesity (BMI > 40)
* Known contraindications to regional anaesthesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of local anaesthetic block. | Over ninety minutes from the start of the study.
  The number of patients in each study arm with altered sensation to cold and pin prick, together with no requirement for opiate analgesia, following surgery was recorded.

SECONDARY OUTCOMES:
Intravenous opiate usage following surgery | 24 hours following surgery
  The usage of intravenous morphine, delivered by a ptient controlled analgesia system, in each group was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Coe, MbChB FRCA, Principal Investigator — Hull and East Yorks NHS Trust
Locations (1):
- Castle Hill Hospital. Castle Road, Cottingham,, Hull, East Yorkshire, United Kingdom